CLINICAL TRIAL: NCT06748300
Title: The Effect of Web-based Breastfeeding Education on Breastfeeding Levels in Adolescent Mothers.
Brief Title: Web-based Breastfeeding Education for Adolescent Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Emine Kurtcan, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Web-Taban
Record Dates: First submitted 2024-12-18; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web taban (Experimental)
  Interventions: Behavioral: web- based education
- face to face (Experimental)
  Interventions: Behavioral: web- based education
- control (No Intervention)

INTERVENTIONS:
Behavioral: web- based education — breastfeeding education
  Other Names: face to face education
  Arms: Web taban; face to face

SUMMARY:
The present study was conducted as a randomized controlled trial to evaluate the effectiveness of web-based and face-to-face breastfeeding education given to primipara adolescent pregnant women. The study was conducted between March 2023 and December 2023 at the University of Health Sciences Van Training and Research Hospital Obstetrics and Gynecology Polyclinics. A total of 135 primipara adolescent pregnant women who met the inclusion criteria were included in the study, including 45 in the Booklet Supported Face-to-Face Breastfeeding Education Program (KİDYEP), 45 in the Web-Based Video Supported Breastfeeding Education Program (WEBVİDEP) and 45 in the control group. Pre-test data were collected in the third trimester by applying socio-demographic data form, breast milk and breastfeeding information form, and breastfeeding self-efficacy short form scale (antenatal form) to the groups. After the pre-test data were collected, a face-to-face breastfeeding education program with a breastfeeding education booklet was administered to the KİDYEP group, and a web-based video-assisted breastfeeding education program was administered to the WEBVİDEP group. Data were collected by applying breast milk and breastfeeding information form, LATCH breastfeeding identification and evaluation scale and breastfeeding self-efficacy short form scale (postnatal version) to the groups at the first (midtest) and sixth (posttest) weeks after delivery. As a result of the present study, the rate of exclusive breastfeeding, the total duration of considering breastfeeding, breast milk and breastfeeding knowledge levels, breastfeeding self-efficacy levels and breastfeeding success of the mothers in the KİDYEP and WEBVİDEP groups were found to be higher than the control group, and both the booklet-supported face-to-face breastfeeding education program and the web-based video-supported breastfeeding education program were found to be similarly effective.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 15 and 19 years
* Being 19 years old and above
* Being literate
* Being primigravida
* Having a single baby (not twins or more)
* Being a volunteer to participate in the study
* Having no health problems for the mother and the baby
* Having a computer, tablet or smart phone and the ability to use it
* Having regular internet access

Exclusion Criteria:

* The mother being 18 years of age or younger
* Being multigravida and/or multiparous
* Having a health problem related to the mother or the baby
* Not having a smart phone or wireless internet during the study period
* Not filling out the survey forms incompletely and not watching videos about hygienic care of the newborn

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
breastfeeding self-efficacy scale | pre-test post-test (approximately seven month)
  breastfeeding self-efficacy scale

CONTACTS AND LOCATIONS:
Locations (1):
- Emine KURTCAN, Van, Lütfen Seçiniz., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No